CLINICAL TRIAL: NCT06181851
Title: Microbiome and Metabolomics Analysis in a Population of Infertile Patients Suffering From Non-obstructive Azospermia and Examination of Their Impact on the Reproductive Potential and Global Health of the Individual
Brief Title: 2015-Metabolomics&Microbiome-infertility
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Andrea Salonia, Professor, IRCCS San Raffaele
Other Study IDs: Metabolomics&microbiome
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Azoospermia, Nonobstructive
MeSH Terms: conditions — Azoospermia, Nonobstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Infertile men: Patients diagnosed with idiopathic non-obstructive azoospermia
  Interventions: Other: Analysis of microbiome and metabolomics
- Fertile men: fertile subjects (pregnancy within 12 months of the start of the research by the couple, according to WHO 2010 criteria)
  Interventions: Other: Analysis of microbiome and metabolomics
- Old fertile men: Subjects known to have been fertile subjects (pregnancy within 12 months of the start of the research by the couple, according to WHO 2010 criteria)
  Interventions: Other: Analysis of microbiome and metabolomics

INTERVENTIONS:
Other: Analysis of microbiome and metabolomics — Analysis of microbiome and metabolomics through the assessment of blood and semen parameters

SUMMARY:
The study aims to carry out a translational analysis of the microbiome and metabolomics in patients suffering from non-obstructive azoospermia, with the aim of investigating prognostic factors predictive of the possible finding of spermatozoa following testicular pulp extraction and differences in blood and seminal level with the fertile population to identify etiopathogenic pathways of this condition.

DETAILED DESCRIPTION:
The study aims to carry out a translational analysis of the microbiome and metabolomics in patients suffering from non-obstructive azoospermia, with the aim of investigating prognostic factors predictive of the possible finding of spermatozoa following testicular pulp extraction and differences in blood and seminal level with the fertile population to identify etiopathogenic pathways of this condition.

Furthermore, the study aims to assess if the blood and seminal alterations of infertile patients have similarities with the same fluids of elderly patients, validating from a metabolomic and microbiomic point of view the hypothesis of premature aging of infertile patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of idiopathic non-obstructive azoospermia
* fertile men (pregnancy within 12 months from the start of the couple's search)
* men known to have been fertile aged between 65 and 75 (pregnancy within 12 months of the couple starting searching)

Exclusion Criteria:

* diagnosis of varicocele
* endocrine alterations
* chromosomal alterations
* known genetic alterations

Ages: 18 Years to 75 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: * diagnosis of idiopathic non-obstructive azoospermia
  * fertile men (pregnancy within 12 months from the start of the couple's search)
  * men known to have been fertile aged between 65 and 75 (pregnancy within 12 months of the couple starting searching)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Prognostic role of the blood and semen samples | Baseline
  Metabolomics and microbiome signature fertile and infertile men predicting possible finding of spermatozoa

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No